CLINICAL TRIAL: NCT07196254
Title: Sandwich Mesh Repair for The Treatment Of Lumbar Incisional Hernia
Brief Title: Lumber Hernia Repair Using Sandwich Mesh Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Yasser Ali Orban, assisstant professor, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sandwich Mesh Repair for The T
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Mesh

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hernia arm represent patients with lumbar abdominal hernia (Experimental): the patient that will undergo sandwich technique repair with onlay and sublay mesh
  Interventions: Procedure: sandwich mesh technique

INTERVENTIONS:
Procedure: sandwich mesh technique — the hernia repair include using double mesh onlay and sublay

SUMMARY:
Lumbar incisional hernia occurs after lumbar incision which is difficult to manage due deficient fascial aponeurosis and a proximity of the bonny boundaries, namely the iliac crest and the last rib. There is a need to evaluate sandwich mesh application, preperitoneal and onlay mesh, in the treatment of lumbar incisional hernia.

ELIGIBILITY:
Inclusion Criteria:

* • Patients older than 18 years old with primary inguinal hernia.

Exclusion Criteria:

* • Pregnancy or patients with bleeding tendency.

  * Complicated hernia.
  * Patients who are not fit for surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
hernia recurrence rate detect by clinical examination and ultrasonography | 6 months starting from the postoperative day 1
  Hernia recurrence is the most critical measure of surgical failure and is a direct indicator of the long-term effectiveness of the repair. A lower recurrence rate demonstrates the superiority of one surgical technique or material over another.

SECONDARY OUTCOMES:
the rate of seroma formation as detected by subcutanous drain | 30 days from postoperative day 1
  the amount if seroma fluid will be estimated in ml as present un surgical subcutanous drain

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig Univeesity Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol